CLINICAL TRIAL: NCT00477711
Title: A Study of Cetuximab(Erbitux) With Cisplatin and Capecitabine(Xeloda)as 1st Line Treatment in the Advanced Gastric Cancer
Acronym: EXTRA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Shen Lin, pro., Peking University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62202-769
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Cancer
Keywords: Cetuximab; cisplatin; capecitabine; first line treatment
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cetuximab; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- C225+Chemotherapy (Experimental)
  Interventions: Drug: cetuximab, cisplatin, capecitabine

INTERVENTIONS:
Drug: cetuximab, cisplatin, capecitabine — Product 1: Cetuximab(Erbitux®) Dosing schedule: 400mg/m2 initial dose and then 250mg/m2 ,weekly dose Mode of administration: intravenously Product 2: capecitabine Dosing schedule: 1000mg/m2 bid, days 1-14, every 3 weeks Mode of administration: orally Product 3: cisplatin Dosing schedule: 80mg/m2, day 1 of every 3 weeks Mode of administration: intravenously

SUMMARY:
The purpose of this study is to investigate whether cetuximab (Erbitux®) with cisplatin and capecitabine (Xeloda) as 1st line treatment in the advanced gastric cancer is effective.

DETAILED DESCRIPTION:
Gastric cancer remains one of the major causes of cancer deaths around the world, especially in Asia. Previous study of ML17032 has proved that XP(capecitabine plus cisplatin)is effective in advanced gastric cancer, with the overall response rate of 41%, the median PFS of 5.6 month. Recently, the EGFR monoclonal antibody of cetuximab has shown to be successful in treating advanced colorectal cancer with or without chemotherapy. Since EGFR also express in gastric cancer, A single arm, open, multicenter phase II study of cetuximab in combination with cisplatin and capecitabine as first line treatment in patient with advanced gastric cancer.If applicable, the value of mutations in k-ras, b-raf, P53, and EGFR copy number to predict the clinical response to cetuximab in advanced gastric cancer patients will also be accessed.Tumor tissue from study patients will be checked for k-ras, b-raf, and P53 mutation by sequencing and for EGFR copy number by chromogenic in situ hybridization. DNA will be extracted from paraffin-embedded samples.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age 18 to 75 years old
* Histologically confirmed gastric adenocarcinoma
* Unresectable recurrent or metastatic disease
* Previous neo-adjuvant or adjuvant treatment for gastric cancer, if applicable, more than 12 months
* Measurable disease according to the RECIST criteria
* Karnofsky performance status ≥60
* Life expectancy of ≥2 month
* No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
* ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)
* Serum albumin level ≥3.0g/dL
* Serum AKP < 2.5 times ULN
* Serum creatinine <1.5mg/dL
* Bilirubin level < 1.5mg/dL
* Serum creatinine <1.5 times ULN
* WBC>3,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl

Exclusion Criteria:

* Brain metastasis (known or suspected)
* Previous systemic therapy for metastatic gastric cancer
* Inability to take oral medication
* Previous EGFR pathway-targeting therapy
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry
* Heart failure, coronary artery disease, myocardial infarction within the last 6 months
* Known allergy to any study treatment
* Pregnancy or lactation period
* Any investigational agent within the past 28 days
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Previous adjuvant therapy with capecitabine+platinum
* Pre-existing neuropathy>grade 1
* Legal incapacity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-03; Primary Completion 2008-12 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Tumor response rate | 1 year

SECONDARY OUTCOMES:
Time to progression Disease control rate Overall survival K-ras, b-raf, p53 gene mutation and EGFR gene copy number vs. tumor response safety | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University, School of oncology, Gastrointestinal Department
Locations (1):
- Peking University,School of Oncology, Gastrointestinal Department, Beijing, China

REFERENCES:
- [Derived] Zhang X, Xu J, Liu H, Yang L, Liang J, Xu N, Bai Y, Wang J, Shen L. Predictive biomarkers for the efficacy of cetuximab combined with cisplatin and capecitabine in advanced gastric or esophagogastric junction adenocarcinoma: a prospective multicenter phase 2 trial. Med Oncol. 2014 Oct;31(10):226. doi: 10.1007/s12032-014-0226-y. Epub 2014 Sep 19. PMID 25234930